CLINICAL TRIAL: NCT05775029
Title: Rapid Sequence Induction Checklist and Its Effect on Compliance to Guidelines and Complications - Follow-up
Brief Title: RSI Observation Follow-up
Status: Active, not recruiting | Type: Observational
Sponsor: Jakob Zeuchner (Other Government)
Responsible Party: Sponsor-Investigator, Jakob Zeuchner, Principal Investigator, Linkoeping University
Organization: Linkoeping University (Other Government)
Other Study IDs: 20220202
Record Dates: First submitted 2022-05-05; First posted 2023-03-20 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: RSI; Rapid Sequence Induction; Complication of Anesthesia; Compliant Behavior
MeSH Terms: conditions — Cooperative Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study group 1: Short term compliance group
- Study group 2: Long term compliance group

SUMMARY:
The purpose of this prospective observational study is to determine if compliance to local guildelines for the RSI procedure, after introduction of a RSI-check list, persists over time (36-60months). Any changes in complication rates will also be evaluated.

DETAILED DESCRIPTION:
A prospective observational study of long-term compliance to local RSI guidelines performed at two hospitals in Region Östergötland County, Sweden. All staff members (specialist anaesthetist, nurse-anaesthetist, resident anaesthetist) performing RSI in adult patients >=18 years of age are eligible for inclusion. Exclusion criteria are refusal to participate, or RSI performed in patients < 18 years old. All members of the staff at the participating centres will be given oral and written information about the study, and consent is implied by completion of the questionnaire.

A standard RSI checklist was introduced in the two hospitals during 2017-2018. The checklist is a 16-item document consisting of statements requiring binary yes/no and "check" type answers and was designed to encourage consistency and completeness in RSI preparations and execution. The statements were based on prior data in literature regarding the RSI procedure. Initial compliance was good when measured at 12 months after implementation of the RSI-checklist and a supporting educational program (Reference 1[Study results]).

The investigators plan to evaluate the long-term compliance to the RSI-checklist. Nurse anaesthetists or anaesthetists attending the patient during RSI will complete a predefined questionnaire about the conduct of RSI and RSI-related complications. The questionnaire will be completed immediately after induction when the patient is stable.

The investigators plan to conduct duplicate measurements in 20% of the observations to test inter-rater variability and to mitigate the risk of bias due to self-reporting.

Primary hypothesis: Compliance to local RSI-guidelines is maintained 36 months after introduction of a pre-RSI checklist.

Secondary hypothesis: Increased compliance to local RSI-guidelines 36 months after introduction of a pre-RSI checklist reduces the frequency of complications

Outcome:

Primary outcome: Compliance to local RSI-guidelines

Compliance categories were defined by consensus of the authors and individual parameters were not weighted. It is measured as a 7-point score, one point for the fulfilment of each seven parameters:

1. 100% FiO2 with FGF >10 L/min for >3 minutes
2. Use of Thiopental or Ketamine
3. Use of Succinylcholine
4. Use of an Orogastric tube
5. Use of a stylet in the endotracheal tube
6. Administration of Sodium Citrate
7. Reverse Trendelenburg or supine patient position

Secondary outcome: Frequency of complications during RSI

Complications are defined as (according to the Swedish Perioperative Registry):

A111: Unexpected difficult airway; > 2 unsuccessful attempts to intubate the patient by an experienced anesthesiologist OR intubation by another, more experienced anesthesiologist than the anesthesiologist responsible for induction.

A126: Hypoxia that requires intervention, e.g. increased fiO2; Hypoxia SpO2 < 90%.

A215: Bradycardia that requires specific pharmacological intervention or change in anesthetic strategy A222: Hypotension that requires unplanned, continuous administration of vasopressor drug.

A514: Dental injury.

ELIGIBILITY:
Inclusion Criteria:

• All staff members (specialist anaesthetist, nurse-anaesthetist, resident anaesthetist) performing RSI in adult patients >=18 years of age.

Exclusion Criteria:

* Refusal of staff member to participate
* RSI performed in patients < 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All staff members (specialist anaesthetist, nurse-anaesthetist, resident) performing RSI in adult patients.
Sampling Method: Probability Sample
Enrollment: 2300 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Compliance to RSI guidelines | 3 years
Change in RSI complication | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Chew, M.D. Ph.D., Study Director — Linkoeping University
Locations (2):
- Sweden (2):
  - Linköping University Hospital, Linköping, Östergötland County
  - Vrinnevisjukhuset, Norrköping, Östergötland County

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stept WJ, Safar P. Rapid induction-intubation for prevention of gastric-content aspiration. Anesth Analg. 1970 Jul-Aug;49(4):633-6. No abstract available. PMID 5534675
- [Background] Zeuchner J, Graf J, Elander L, Frisk J, Fredrikson M, Chew MS. Introduction of a rapid sequence induction checklist and its effect on compliance to guidelines and complications. Acta Anaesthesiol Scand. 2021 Oct;65(9):1205-1212. doi: 10.1111/aas.13947. Epub 2021 Jul 26. PMID 34173228
- [Background] Klucka J, Kosinova M, Zacharowski K, De Hert S, Kratochvil M, Toukalkova M, Stoudek R, Zelinkova H, Stourac P. Rapid sequence induction: An international survey. Eur J Anaesthesiol. 2020 Jun;37(6):435-442. doi: 10.1097/EJA.0000000000001194. PMID 32221099
- [Background] Jensen AG, Callesen T, Hagemo JS, Hreinsson K, Lund V, Nordmark J; Clinical Practice Committee of the Scandinavian Society of Anaesthesiology and Intensive Care Medicine. Scandinavian clinical practice guidelines on general anaesthesia for emergency situations. Acta Anaesthesiol Scand. 2010 Sep;54(8):922-50. doi: 10.1111/j.1399-6576.2010.02277.x. PMID 20701596
- [Background] Koerber JP, Roberts GE, Whitaker R, Thorpe CM. Variation in rapid sequence induction techniques: current practice in Wales. Anaesthesia. 2009 Jan;64(1):54-9. doi: 10.1111/j.1365-2044.2008.05681.x. PMID 19087008
- [Background] Pugel AE, Simianu VV, Flum DR, Patchen Dellinger E. Use of the surgical safety checklist to improve communication and reduce complications. J Infect Public Health. 2015 May-Jun;8(3):219-25. doi: 10.1016/j.jiph.2015.01.001. Epub 2015 Feb 26. PMID 25731674
- [Background] Sullivan A, Elshenawy S, Ades A, Sawyer T. Acquiring and Maintaining Technical Skills Using Simulation: Initial, Maintenance, Booster, and Refresher Training. Cureus. 2019 Sep 23;11(9):e5729. doi: 10.7759/cureus.5729. PMID 31723493